CLINICAL TRIAL: NCT03467750
Title: Ketorolac as a Strategy for Reducing Post-operative Opioid Requirements in Children With Obstructive Sleep Apnea Undergoing Adenotonsillectomy: a Randomized Controlled Trial
Brief Title: Effect of Ketorolac on Post Adenotonsillectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Laura Gilbertson, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00097738
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Adenotonsillectomy; Opioids; Post-surgical pain; Anesthesiology; Pediatrics
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Standard of Care; Sevoflurane; Propofol; Calcium Dobesilate; Dexmedetomidine; Ondansetron; Morphine

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The PACU nurses will be blinded to ketorolac administration, but will be informed of all other medications given. The PACU nurses will evaluate the patients using FLACC scores at 10 minutes post-op, 20 minutes post-op and at time of PACU discharge. Morphine will be administered to obtain a FLACC score of less than 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketorolac (Experimental): Participants randomized to the ketorolac group will receive 0.5mg/kg IV at the end of the adenotonsillectomy procedure, once hemostasis has been achieved
  Interventions: Drug: Ketorolac; Drug: Standard of Care
- Standard of Care (Active Comparator): Participants randomized to this group will receive the pain management standard of care for the adenotonsillectomy procedure.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Ketorolac — Patients in this group will receive 0.5mg/kg of ketorolac, administered intravenously.
  Other Names: Toradol
  Arms: Ketorolac
Drug: Standard of Care — All patients will undergo inhalational induction with nitrous oxide and sevoflurane. After intravenous (IV) placement, 1-3mg/kg of propofol and 1mcg/kg of fentanyl will be administered. After induction, 0.5mg/kg of dexamethasone and an IV infusion of 15mg/kg of acetaminophen will be administered. During surgery, 0.5mcg/kg of dexmedetomidine and 0.1mg/kg ondansetron will be given.
  A rescue dose of 0.5-1mcg/kg of IV Fentanyl will be available for use at the end of the procedure. The decision to administer will be left to the discretion of the attending anesthesiologist. The choice to give this will be made based on variables including patient's condition and a 20% increase in the heart rate and blood pressure.
  The PACU nurses, who will be blinded to ketorolac administration, will evaluate the patients using FLACC scores. For patients with a FLACC score of 6-10, morphine 0.05mg/kg will be administered. For patients with FLACC scores of 3-5, morphine 0.025mg/kg will be administered.
  Other Names: Sojourn; Ultane; Diprivan; Decadron; Precedex; Zofran; Morphine

SUMMARY:
This randomized prospective study aims to determine the effect of ketorolac on the total dose of morphine required to achieve postoperative analgesia in children with obstructive sleep apnea (OSA) undergoing adenotonsillectomy. Participants will be randomly assigned to a study group where they will receive ketorolac in addition to the standard of care treatment or will receive only the standard of care pain management. The researchers hypothesize that by administering ketorolac at the end of the procedure once hemostasis has been achieved, it will be possible to decrease the amount of morphine administered in the post-anesthesia care unit (PACU). This study aims to provide a more comprehensive understanding of the efficacy and safety of the current standard post-operative analgesic regimen employed at the study institution, in which opioid analgesia currently plays a prominent role.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) as an indication for adenotonsillectomy has increased significantly over the past ten years, and now has surpassed recurrent tonsillitis as the most common indication for this procedure. Opioids continue to be the most commonly administered pain medication for these procedures. Studies have shown that patients with OSA have significantly increased sensitivity to opioids that results in post-operative respiratory depression and apnea when administered via standard opioid dosing protocols. Children with OSA were shown to have a nearly fivefold increase in the odds of developing respiratory complications when compared to their counterparts with tonsillitis. Ketorolac possesses similar efficacy to morphine without the problematic complications of respiratory depression, nausea and vomiting, which are commonly seen post-adenotonsillectomy. Importantly, when combined with opioids, ketorolac is opioid-sparing. This synergistic effect means that a similar level of analgesia is achieved using a lower dose of opioid. However, there continues to be concern about using ketorolac due to the potential risk of post-operative bleeding from anti-platelet activity.

This randomized, prospective study aims to determine the effect of ketorolac on the total dose of morphine required to achieve postoperative analgesia in children with OSA undergoing adenotonsillectomy. Participants will be randomly assigned to receive ketorolac or to not receive ketorolac. The post-anesthesia care unit (PACU) nurses, who will be blinded to ketorolac administration, will evaluate the patients using the Face, Legs, Activity, Cry, Consolability (FLACC) scale scores at 10 minutes post-op, 20 minutes post-op and at time of PACU discharge. For patients with a FLACC score of 6-10, morphine (0.05mg/kg) will be administered. For patients with FLACC scores of 3-5, morphine (0.025mg/kg) will be administered. The total amount of opioid required to obtain a FLACC score of less than 3 will be evaluated as the primary outcome. The secondary outcomes to be evaluated will be PACU FLACC scores, time required in PACU, incidence of post-tonsillectomy bleeding and total pain medications administered during hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sleep disordered breathing or obstructive sleep apnea
* Children undergoing elective tonsillectomy or adenotonsillectomy at Children's Healthcare of Atlanta Egleston location
* Parent or legal guardian willing to participate, and able to understand and sign the provided informed consent

Exclusion Criteria:

* Known coagulation defect
* Patients on longstanding NSAID therapy
* Known renal impairment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gilbertson, MD, Principal Investigator — Emory University
Locations (1):
- Childrens Healthcare of Atlanta, Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta at Egleston in Atlanta, Georgia, USA. Participant enrollment began July 19, 2018 and the final study assessment occurred on August 22, 2023.
Groups:
- Ketorolac: Participants randomized to the ketorolac group received 0.5mg/kg IV at the end of the adenotonsillectomy procedure, once hemostasis was achieved.
  Ketorolac: Patients in this group received 0.5mg/kg of ketorolac, administered intravenously.
  Standard of Care: All patients underwent inhalational induction with nitrous oxide and sevoflurane. After intravenous (IV) placement, 1-3mg/kg of propofol and 1mcg/kg of fentanyl were administered. After induction, 0.5mg/kg of dexamethasone and an IV infusion of 15mg/kg of acetaminophen were administered. During surgery, 0.5mcg/kg of dexmedetomidine and 0.1mg/kg ondansetron were given.
  A rescue dose of 0.5-1mcg/kg of IV Fentanyl was available for use at the end of the procedure. The decision to administer was left to the discretion of the attending anesthesiologist. The choice to give this was made based on variables including patient's condition and a 20% increase in the heart rate and blood pressure.
  The PACU nurses, who were blinded to ketorolac administration, evaluated the patients using FLACC scores. For patients with a FLACC score of 6-10, morphine 0.05mg/kg was administered. For patients with FLACC scores of 3-5, morphine 0.025mg/kg was administered.
- Standard of Care: Participants randomized to this group received the pain management standard of care for the adenotonsillectomy procedure.
  Standard of Care: All patients underwent inhalational induction with nitrous oxide and sevoflurane. After intravenous (IV) placement, 1-3mg/kg of propofol and 1mcg/kg of fentanyl were administered. After induction, 0.5mg/kg of dexamethasone and an IV infusion of 15mg/kg of acetaminophen were administered. During surgery, 0.5mcg/kg of dexmedetomidine and 0.1mg/kg ondansetron were given.
  A rescue dose of 0.5-1mcg/kg of IV Fentanyl was available for use at the end of the procedure. The decision to administer was left to the discretion of the attending anesthesiologist. The choice to give this was made based on variables including patient's condition and a 20% increase in the heart rate and blood pressure.
  The PACU nurses, who were blinded to ketorolac administration, evaluated the patients using FLACC scores. For patients with a FLACC score of 6-10, morphine 0.05mg/kg was administered. For patients with FLACC scores of 3-5, morphine 0.025mg/kg was administered.
Period: Overall Study
Arm/Group | Ketorolac | Standard of Care
Started | 30 | 33
Completed | 28 | 31
Not Completed | 2 | 2
Not completed — Surgery canceled | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketorolac: Participants randomized to the ketorolac group received 0.5mg/kg IV at the end of the adenotonsillectomy procedure, once hemostasis was achieved.
- Standard of Care: Participants randomized to this group received the pain management standard of care for the adenotonsillectomy procedure.
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Standard of Care | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.43 (3.20) | 4.36 (2.91) | 4.40 (3.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 30
  Male | 19 | 14 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 20 | 34
  White | 16 | 10 | 26
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Post-Anesthesia Care Unit (PACU) Morphine Requirements
Description: The total postoperative morphine dosage required to achieve analgesia (defined as a Face, Legs, Activity, Cry, Consolability (FLACC) Scale score of less than 3) in children with obstructive sleep apnea undergoing adenotonsillectomy was compared between study arms to examine the effect of ketorolac administration.
Time Frame: Until PACU discharge (up to 261 minutes)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Ketorolac | Standard of Care
Number analyzed (Participants) | 28 | 31
mg/kg | 0.033 (0.034) | 0.058 (0.096)

2. Secondary Outcome: Face, Legs, Activity, Cry, Consolability (FLACC) Scale Score
Description: Post-Anesthesia Care Unit (PACU) nurses evaluated the patients using Face, Legs, Activity, Cry, Consolability (FLACC) Scale scores at 10 minutes post-op, 20 minutes post-op and at time of PACU discharge. Each category is scored as 0 (no indication of pain), 1 (indication of moderate pain), or 2 (visibly experiencing severe pain). Total scores range from 0 to 10, with higher scores indicating more pain.
Time Frame: 10 minutes post-op, 20 minutes post-op, PACU discharge (up to 261 minutes)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketorolac | Standard of Care
Number analyzed (Participants) | 28 | 31
score on a scale
  10 minutes post-op | 1.74 (2.80) | 2.87 (3.86)
  20 minutes post-op | 2.37 (3.13) | 3.23 (3.67)
  PACU discharge | 0.85 (1.13) | 0.77 (1.15)

3. Secondary Outcome: Post-Anesthesia Care Unit (PACU) Recovery Time
Description: The duration of time that a participant was in the Post-Anesthesia Care Unit (PACU), following surgery, measured in minutes.
Time Frame: Until PACU discharge (up to 261 minutes)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ketorolac | Standard of Care
Number analyzed (Participants) | 28 | 31
minutes | 63.4 (39.9) | 49.7 (12.2)

4. Secondary Outcome: Number of Participants With Post-Tonsillectomy Bleeding
Description: Participants were monitored via medical chart review for post-tonsillectomy bleeding.
Time Frame: Up to 14 days after surgery
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac | Standard of Care
Number analyzed (Participants) | 28 | 31
Participants | 1 | 2

5. Secondary Outcome: Pain Medication Administration
Description: The total amount of pain medications administered during hospitalization was examined.
Time Frame: Surgery through hospital discharge (up to post-operative day 2)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Error); unit: Morphine Equivalents in mg/kg
Arm/Group | Ketorolac | Standard of Care
Number analyzed (Participants) | 28 | 31
Morphine Equivalents in mg/kg | 0.017 (0.04) | 0.040 (0.093)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected among participants who completed the surgery, beginning at the time of consent and continued through the final assessment at complete recovery, up to 14 days after surgery.
Description: Post-tonsillectomy bleeding requiring surgery is a known risk of tonsillectomy and is not considered to be a serious adverse event in this study.
Arm/Group | Ketorolac | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 1/29 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=29) | Standard of Care (N=32)
Post-operative bleeding requiring surgery (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03467750/Prot_SAP_000.pdf